CLINICAL TRIAL: NCT01624493
Title: Phase I/II BNC105P Combination Study in Partially Platinum Sensitive Ovarian Cancer Patients in First or Second Relapse
Brief Title: BNC105P Combination Study in Partially Platinum Sensitive Ovarian Cancer Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Phase I was conducted Australia. Phase II not conducted and no US pts enrolled.
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: University of Sydney (Other); Australia New Zealand Gynaecological Oncology Group (Other); Bionomics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GYN12-154 / ANZGOG-1103
Record Dates: First submitted 2012-06-15; First posted 2012-06-20 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Ovarian Cancer
Keywords: Vascular Disrupting Agents; BNC105P; Partially platinum sensitive
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Gemcitabine; BNC 105P

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase II Arm A (Experimental): Phase II Arm A will randomize patients to treatment regimen of carboplatin and gemcitabine without BNC105P
  Interventions: Drug: Carboplatin; Drug: Gemcitabine
- Phase II Arm B (Experimental): Phase II Arm B will randomize patients to treatment regimen of carboplatin and gemcitabine and will include BNC105P
  Interventions: Drug: Carboplatin; Drug: Gemcitabine; Drug: BNC105P

INTERVENTIONS:
Drug: Carboplatin — Carboplatin AUC4 on day 1 of 21-day cycle, for a maximum of 6 cycles.
  Arms: Phase II Arm A
Drug: Gemcitabine — Gemcitabine escalations 800 and 1000 mg/m2 (as determined in phase I) on days 1 and 8 of a 21 day cycle, for a maximum of 6 cycles.
  Arms: Phase II Arm A
Drug: Carboplatin — Carboplatin AUC 4 on day 1 of a 21 day cycle, for a maximum of 6 cycles.
  Arms: Phase II Arm B
Drug: Gemcitabine — Gemcitabine 800 or 1000 mg/m2 (as determined in phase I) on days 1 and day 8 of 21-day cycle, for a maximum of 6 cycles.
  Arms: Phase II Arm B
Drug: BNC105P — BNC105P as determined in phase I, on days 2 and 9 of a 21 day cycle for a maximum of 6 cycles, followed by single agent maintenance BNC105P 16 mg/m2 for a maximum of 6 additional cycles.
  Arms: Phase II Arm B

SUMMARY:
This phase I/II trial will determine the recommended dose and activity of BNC105P for patients with partially platinum sensitive ovarian cancer in first or second relapse.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

BNC105P is a novel vascular disrupting agent (VDA) with promising preclinical activity combined with platinum or gemcitabine. The results of standard chemotherapy with carboplatin and gemcitabine for ovarian cancer relapsing within 12 months of an initial platinum-based regimen require improvement. This trial will determine the recommended dose and activity of BNC105P administered with carboplatin and gemcitabine.

PHASE I:

This trial uses a standard 3+3 design for allocating participants to a starting dose level in Phase I.

If dose level 1 is deemed to have acceptable toxicity then dose levels 2a and 2b can be opened at the same time. Dose level 3 will only open if both dose levels 2a and 2b are deemed to have acceptable toxicity.

The underlying assumptions for determining the recommended doses for the triple combination of carboplatin, gemcitabine and BNC105P are that the likely minimum doses required of each agent are carboplatin AUC 4, gemcitabine 800 mg/m2 and BNC105P 12 mg/m2. This corresponds to dose level 1.

PHASE II 1:1 RANDOMIZATION:

Carboplatin AUC 4 on day 1, gemcitabine 800 or 1000 mg/m2 on days 1 and 8 of a 21 day cycle for a maximum of 6 cycles.

OR

Carboplatin AUC 4 on day 1, gemcitabine 800 or 1000 mg/m2 on days 1 and day 8 with dose of BNC105P as determined in phase I, on days 2 and 9 of a 21 day cycle for a maximum of 6 cycles, followed by single agent maintenance BNC105P 16 mg/m2 for a maximum of 6 additional cycles

Minimum follow up for 12 months

ECOG Performance Status for Phase I: 0-1; ECOG Performance Status for Phase II: 0-2

Life Expectancy: Less than 12 weeks

Hematopoietic (both phases):

* Platelet count ≥ 100 x 109/L
* ANC ≥ 1.5 x 109/L
* Haemoglobin > 9g/dl (can be post transfusion)
* INR ≤ 1.5 x ULN

Hepatic (both phases):

* Total Bilirubin ≤ 1.5 x the upper limit of normal (ULN)
* ALT ≤ 2.5 x ULN

Renal (both phases):

* Creatinine clearance ≥ 55 mL/min according to Cockcroft Gault formula
* If Calculated GFR is 50 - 54 mL/min an isotopic GFR may be performed. If the isotopic GFR is > 55ml/min, the patient will be eligible for the study but the calculated GFR will be used for dose calculation.

Cardiovascular (both phases):

* Normal left ventricular ejection fraction (LVEF), i.e. ≥ 50% on Gated Heart Pool Scan, or fractional shortening on echocardiogram ≥ institutional LLN performed within 2 months prior to randomisation
* Corrected QTc < 470 msec on ECG performed within 4 weeks prior to randomisation.

ELIGIBILITY:
Inclusion Criteria for Phase I Only:

* Histologically or cytologically proven diagnosis of epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer, including all histological subtypes and carcinosarcoma.

Inclusion Criteria for Phase II Only:

* Histologically proven diagnosis of epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer.
* Progression-free interval between 4 to 9 months after first line chemotherapy or 4 to 12 months after second-line chemotherapy with a platinum (cisplatin or carboplatin) based regimen.
* Subjects must have progressed (based on GCIG CA125 and/or RECIST criteria) after last platinum based regimen.
* Subjects must be assessable for response based on GCIG CA125 and/or RECIST criteria.
* Subjects with clinically evident ascites and/or pleural effusions must be assessable by RECIST.
* Study treatment both planned and able to start within 7 days of randomisation

Exclusion Criteria for Phases I and II:

* Non-epithelial ovarian cancer and ovarian tumours of low malignant potential (borderline tumours)
* More than two prior chemotherapy regimens for ovarian cancer (excluding hormonal therapy or biologic agents).
* Any prior chemotherapy for other cancers, but >10 years permitted for phase II only, except for high dose chemotherapy/autologous or allogeneic transplantation
* Chemotherapy within 20 days prior to registration.
* Hormonal therapy or biologic therapy within 28 days prior to registration
* Concurrent treatment with any experimental drugs or other anti-cancer therapy.
* Concurrent treatment with clopidogrel, ticlopidine, persantin and other antiplatelet agents
* Radiotherapy within 21 days prior to registration, or to greater than 15% of the bone marrow.
* Persistent toxic effects of previous chemotherapy of greater than Grade 1 severity (CTCAE v 4, appendix 8)
* Known brain or leptomeningeal disease (baseline CT brain or MRI is only required if there is clinical suspicion of central nervous system involvement).
* Subjects with other invasive malignancies who had (or have) any evidence of another cancer present within the last 3 years, with the exception of early stage non-melanoma skin cancer, carcinoma in situ of cervix, and synchronous endometrial cancer (stage 1 G1,2)
* Untreated and/or uncontrolled cardiovascular conditions and/or symptomatic cardiac dysfunction (unstable angina, congestive cardiac failure, myocardial infarction) within the previous year, or cardiac ventricular arrhythmias requiring medication, or history of 2nd or 3rd degree atrioventricular conduction defects.
* Cerebrovascular accident or transient ischemic attack within 6 months prior to registration.
* Poorly controlled hypertension: systolic BP >150 or diastolic BP >100 mmHg. Antihypertensive medications are permitted but BP must be ≤150 systolic and ≤100 diastolic on 2 readings separated by at least 24 hours.
* Deep vein thrombosis, pulmonary embolism, within 6 months of registration or arterial thrombosis, or arterial embolism within 12 months prior to registration.
* Receiving full dose, therapeutic anti-coagulation with warfarin, related oral anti-coagulants or unfractionated or low molecular weight heparin. Low dose heparin given for prophylaxis, and aspirin at a dose ≤ 325 mg/day is acceptable.
* Significant infection including active hepatitis B, hepatitis C with abnormal liver function tests, or HIV. Testing for these is not mandatory. Screening for Hepatitis B should be as per institutional policy. Patients known to be Hep B surface antigen positive will be not be eligible even if on antiviral treatment.
* Serious medical or psychiatric conditions which might prevent management according to the protocol.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomisation
* Pregnancy, lactation, or inadequate contraception. Women must be post menopausal or sterile, or use two reliable means of contraception. Women of childbearing potential must have a pregnancy test taken and proven negative within 7 days prior to registration.
* Life expectancy of less than 12 weeks.

Exclusion Criteria for Phase II only:

* Carcinosarcoma and mucinous carcinoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Phase I: Determine Maximum Tolerated Dose for Patients | 12 months
  To determine the recommended dose of BNC105P given with gemcitabine and carboplatin (maximum dose of BNC105P with no more than 1 DLT in 6 phase I participants)
Phase II: Determine Objective Response Rate in Patients | 12 months
  To determine the objective response rate (ORR) in those with evaluable disease (ORR = CR, PR according to RECIST 1.1 and/or GCIG CA125 criteria) (percentage of those with measurable disease achieving CR or PR according to RECIST 1.1 and/or GCIG CA125 criteria)

SECONDARY OUTCOMES:
Progression Free and Overall Survival Distribution | 12 months
  To determine the progression free and overall survival distribution rates in this patient population
Patient Side Effects and Tolerability | 12 months
  To determine the adverse event rates (Numbers (%) with G2-5 AE (NCI CTCAE v4.0)
Patient Quality of Life Benefits | 12 months
  To determine the effects on aspects of health related quality of life (HRQL measured with FOSI and MOST), including symptom benefit (Numbers (%) with significant symptom benefit)
Assessment of BNC105P Pharmacokinetics to Determine Interaction with Carboplatin and Gemcitabine | 12 months
  Plasma will be collected to assess BNC105P pharmacokinetics on days 2 and 9 of cycle 1 only. Results will be compared with data from previous trials of BNC105P to determine their consistency and to establish if there is any major interaction with carboplatin and gemcitabine.
Association of Biomarkers, Predictions and Outcomes | 12 months
  To determine the associations between baseline biomarkers, ORR, PFS, OS and AE

CONTACTS AND LOCATIONS:
Overall Officials: Danny Rischin, Professor, Study Chair — University of Sydney; Daniela Matei, M.D., Principal Investigator — Hoosier Cancer Research Network
Locations (6):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
- Australia (3):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Christchurch Hospital, Christchurch, Canterbury, New Zealand

REFERENCES:
- [Background] Danny Rischin, Daniela Matei, Jeffrey C. Goh, Michelle Margaret Vaughan, Philip James Beale, Meaghan Elizabeth Tenney, Julie Martyn, Dirkje Willemien Sommeijer, Jose Luis Iglesias, David C. Bibby, Jeremy Simpson, Elizabeth E. Doolin, Corinne E. Williams, Martin R. Stockler. A phase I/II study of the vascular disrupting agent BNC105P in combination with gemcitabine-carboplatin in partially platinum-sensitive ovarian cancer patients in first or second relapse: An international collaborative group trial of ANZGOG and HOG. J Clin Oncol 31, 2013 (suppl; abstr TPS5612) http://abstracts2.asco.org/AbstView_132_108013.html
- [Background] Danny Rischin, Philip James Beale, Emma Caroline Rossi, Jeffrey C. Goh, Michelle Margaret Vaughan, Meaghan Elizabeth Tenney, Julie Martyn, Dirkje Willemien Sommeijer, Jose Luis Iglesias, Gabriel Kremmidiotis, Jeremy Andrew Simpson, Elizabeth E. Doolin, Tina C. Lavranos, Annabell F. Leske, Anne-Sophie Veillard, Martin R. Stockler, ANZGOG and HOG. A phase I study of the vascular-disrupting agent BNC105P in combination with gemcitabine-carboplatin in platinum-sensitive ovarian cancer patients in first or second relapse. J Clin Oncol 32:5s, 2014 (suppl; abstr 5524^). ACTRN12612000522819
- See also: Hoosier Oncology Group Website — http://www.hoosieroncologygroup.org